CLINICAL TRIAL: NCT05598086
Title: Anti-fibrinolytic and Anti-inflammatory Effects of Local Infiltration of Tranexamic Acid in the Post-operation of Displaced Intra-articular Calcaneal Fractures: a Randomized Controlled Study
Brief Title: Anti-fibrinolytic and Anti-inflammatory Effects of Local Infiltration of Tranexamic Acid in Patients With Calcaneal Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TXA01
Record Dates: First submitted 2022-10-22; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Tranexamic Acid; Fibrinolysis; Inflammatory; Fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA group (Experimental): Postoperative 1g TXA was infiltrated locally around the incision immediately for patients in TXA group.
  Interventions: Drug: Tranexamic acid
- Normal saline group (Placebo Comparator): 1 g 0.9% saline was infiltrated locally around the incision immediately after surgery for patients in normal saline group.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — local infiltration of TXA or normal saline in the post-operation would
  Other Names: Normal saline

SUMMARY:
Background. Consensus is lacking regarding the use of tranexamic acid (TXA) in calcaneal fracture surgery. This study aims to investigate the hypothesis that local infiltration of TXA in the post-operation would maintain hemoglobin (Hb) level, reduce incision drainage volume and risk of infection in patients with displaced intra-articular calcaneal fractures. Methods. A total of 120 patients with displaced intra-articular calcaneal fractures who received extensible lateral L-shaped approach were included in this trial and equally randomized to receive one single dose of 1g TXA or 1g normal saline after closing incision. The demographic data and fracture characteristics, intra-operative indicators, laboratory tests and Visual Analogue Scale (VAS) scores, incision drainage volume, and incision-related complications were collected and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with age of eighteen years or older;
* diagnosis of closed and unilateral displaced intra-articular calcaneal fracture;
* agreement to receive one of the two treatment strategies;
* agreement to participate in regular follow-up after surgery

Exclusion Criteria:

* open calcaneal fractures;
* polytrauma of the ipsilateral lower limb;
* systemic inflammatory or infectious diseases;
* previous history of calcaneal fracture or bone tumor;
* allergies to drugs used, or refused to accept the specified treatment strategy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Incision drain output (mL) | 2 days
  Incision drain output of post-operative day 1 and 2
Outcomes of laboratory test | 4 days
  White blood cell (10^9/L)
Outcomes of laboratory test | 4 days
  Neutrophil count (10^9/L)
Outcomes of laboratory test | 4 days
  Hemoglobin (g/L)

SECONDARY OUTCOMES:
Incidence of surgical related complications | 30 days
  Complications included oozing of the blood, hematoma, or deep infection etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Medical University Third Hospital, Shijiazhuang, Hebei, China